CLINICAL TRIAL: NCT00644813
Title: Clinical Outcomes Following Glenoid Neck Fracture as Correlated With Quantitative Assessment of Osseous Injury
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: H-26863
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Scapula Fracture; Glenoid; Fracture
Keywords: Scapula fracture involving glenoid neck; Forelimb dysfunction
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Scapular with glenoid neck fractures: Collect outcome and radiological data on patients with scapular fractures involving the glenoid neck (bone joining the shoulder joint and the scapular body) for a period of 1 year.
  Interventions: Other: Scapular with glenoid neck fractures

INTERVENTIONS:
Other: Scapular with glenoid neck fractures

SUMMARY:
A significant subset of patients with scapula fractures also involves the glenoid neck (bone joining the shoulder joint the scapular body). There is little evidence pertaining to the best treatment or precise definition of these lesions. This study will be designed as a prospective, non-randomized cohort study that will collect outcome and radiological data on patients who have sustained a fracture of the glenoid neck (bone joining the shoulder joint the scapular body) for a period of 1 year. All patients who have sustained extraarticular scapula fractures (any fracture not involving the glenoid surface) will be considered. Information will be collected with respect to the radiographic characteristics of osseous injuries as well as functional outcome over time.

DETAILED DESCRIPTION:
Extraarticular fractures (fracture not involving the glenoid articular surface) of the scapula (shoulder blade) have been traditionally managed nonoperatively. The logic for this course of treatment was based on the healing potential of the extensive muscular envelop of the scapula, the inherent mobility of the shoulder joint, and the difficulty in objectively assessing the degree of injury given its irregular osseous architecture.

Scapular fractures specifically involving the glenoid neck have the potential to significantly change the geometry of glenohumeral joint (shoulder joint) as well as affect the actions of muscles and nerves that act across it. Although most reports indicate patients sustaining glenoid neck fractures did well following nonoperative treatment, there was little use of validated outcome measures. Additionally, the context of severe trauma may have lead to an underestimation of functional recovery.

Advances in imaging technology combined with the evolution of internal fixation techniques have resulted in sporadic attempts at fixation of glenoid neck fractures, usually when they occurred in concert with bony injury to other members of the shoulder girdle, as in the "floating shoulder". However, in the absence of a universal canon of radiograph measurements, there are no current recommendations for operative versus non-operative management based on the characteristics of osseous injury as correlated with probable clinical outcome. Moreover, the common assertion that nonoperative management of scapular fractures leads to adequate functional outcome has not been rigorously examined in a prospective fashion, despite this being the standard of care nationally.

Recent evidence suggests that nonoperative treatment may lead to significant decreases in strength and forelimb function despite the fact that the standard of care for the vast majority of these injuries does not involve surgery or reduction. The same may be true of glenoid neck fractures, as significant shortening or angulation of this metaphyseal isthmus may have a detrimental effect on the functional geometry of the glenohumeral (shoulder) joint. If so, surgical management may be indicated to restore a more physiologic geometry to the joint, and thereby give the best chance of recovery to a pre-injury level of function. It is our hope that these correlates of measurements and outcome will help codify an a priori set of radiograph evaluation criteria to help guide decisions for surgical versus non-operative management of glenoid neck fractures. The purpose of the study is to: 1) define the degree of forelimb dysfunction brought about by this specific injury and 2) the magnitude of osseous injury to the glenoid neck that can be tolerated before functional outcome is unacceptably impeded.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 and 65+
* Extraarticular scapular fractures Scapular fracture is isolated or in concert with nondisplaced ipsilateral fractures of the clavicle, coracoid or acromion or has a clavicle fracture been operatively reduced or fixed?
* Patient is free of preexisting neuromuscular or psychiatric dysfunction
* Patient is free of previous upper extremity injury that would impede objective functional outcome evaluation
* Patient received a CT scan as part of their initial clinical care
* Patient is English speaking
* Patient is signed the informed consent form

Exclusion Criteria:

* Preexisting upper extremity injury or neuromuscular condition
* Displaced fractures of the acromion, clavicle, or coracoid
* Concomitant injury to the forelimb
* Patients mentally or physically unable to perform the function evaluation
* Patients unwilling or unable to follow up for 1 year
* Patients with poor propensity to follow up; drug, alcohol issues, etc.
* Non English speaking patients
* Patients currently or pending incarceration in prison

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gender: Both Age: Adult (18-64 yrs), Geriatric (65+ yrs) Ethnicity: All Ethnic Groups Languages: English Groups to be recruited will include: Patients only
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2008-03; Primary Completion 2017-12 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Displaced Fractures | 12 months, 24 months (optional)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tornetta, MD, Principal Investigator — Boston University / Boston Medical Center
Locations (13):
- United States (12):
  - Indiana University, Indianapolis, Indiana
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan Health system, Ann Arbor, Michigan
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Orthopaedic associates of Michigan, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Charlotte Medical Center, Charlotte, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Orthopaedic Specialty Associates - Fort Worth, Fort Worth, Texas
  - University of Utah, Salt Lake City, Utah
- QEII Health Science Center, Halifax, Canada